CLINICAL TRIAL: NCT00694304
Title: A Long-term, Open-label, Flexible-dose, Extension Study Evaluating the Safety and Tolerability of [Vortioxetine] Lu AA21004 in Patients With Major Depressive Disorder
Brief Title: Open-label Safety Extension Study of 2.5, 5 and 10 mg of Vortioxetine (Lu AA21004) in Long-term Treatment of Major Depressive Disorder in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11984B; EudraCT 2007-004992-21 (Registry Identifier: EudraCT)
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Long-term; Safety; Open-label
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vortioxetine (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)

INTERVENTIONS:
Drug: Vortioxetine (Lu AA21004) — 2.5, 5, or 10 mg/day; tablets; orally
  Other Names: Brintellix

SUMMARY:
The purpose of the study is to evaluate long-term safety and tolerability of Vortioxetine over a period of 52 weeks in patients with Major Depressive Disorder (MDD) having completed 8-week acute treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patients who completed 8-week short-term treatment study for Major Depressive Episode, NCT00635219 / 11984A

Exclusion Criteria:

* Any current psychiatric disorder other than MDD as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Ed., Text revision (DSM-IV TR)
* Female patients of childbearing potential who are not using effective contraception
* Use of any psychoactive medication

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Result] Baldwin DS, Hansen T, Florea I. Vortioxetine (Lu AA21004) in the long-term open-label treatment of major depressive disorder. Curr Med Res Opin. 2012 Oct;28(10):1717-24. doi: 10.1185/03007995.2012.725035. Epub 2012 Sep 17. PMID 22978748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients eligible to participate in Study 11984B were patients who had completed lead-in Study NCT00635219 / 11984A immediately prior to inclusion into Study 11984B.
Pre-assignment Details: The study consisted of a 52-week open-label period and a 4-week Safety Follow-up Period.
Groups:
- Vortioxetine 2.5, 5, or 10 mg/Day: tablets; orally
Period: Overall Study
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Started | 535
Completed | 328
Not Completed | 207
Not completed — Adverse Event | 42
Not completed — Lack of Efficacy | 35
Not completed — Non-compliance With Study Product | 16
Not completed — Protocol Violation | 6
Not completed — Withdrawal of Consent | 61
Not completed — Lost to Follow-up | 15
Not completed — Administrative or Other Reasons | 32

BASELINE CHARACTERISTICS:
Population: Age and Sex: all-patients-treated set (APTS) - all patients who took at least one dose of Vortioxetine after Baseline; MADRS, HAM-D-24, HAM-A, CGI-S and SDS: full-analysis set (FAS) - all patients in the APTS who had at least one valid post-Baseline assessment of the MADRS total score.
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Number analyzed (Participants) | 535
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 366
  Male | 169
MADRS [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
  units on a scale | 13.5 (8.7)
HAM-D-24 [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Scale - 24 Items (HAM-D-24) measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 76. The higher the score, the more severe.
  units on a scale | 13.4 (8.7)
HAM-A [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
  units on a scale | 11.0 (7.2)
CGI-S [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
  units on a scale | 2.7 (1.2)
SDS [Mean (Standard Deviation); unit: units on a scale] — The Sheehan Disability Scale (SDS) comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). The higher the score, the more severe.
  units on a scale | 12.42 (8.13)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs)
Time Frame: Baseline to end of the 4-week safety follow-up period
Population: APTS
Measure: Number; unit: participants
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Number analyzed (Participants) | 535
participants
  Patients With AEs | 391
  Patients With SAEs | 18
  Patients With AEs Leading to Withdrawal | 42

2. Primary Outcome: Percentage of Patients Who Withdrew Due to Intolerance to Treatment
Time Frame: Baseline to Week 52
Population: APTS
Measure: Number; unit: percentage of patients
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Number analyzed (Participants) | 535
percentage of patients | 7.7

3. Secondary Outcome: Change From Baseline in MADRS Total Score After 52 Weeks of Treatment
Description: The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
Time Frame: Baseline and Week 52
Population: FAS; observed cases (OC)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Number analyzed (Participants) | 329
units on a scale | -7.35 (8.21)

4. Secondary Outcome: Change From Baseline in HAM-D-24 Total Score After 52 Weeks of Treatment
Description: The Hamilton Depression Scale - 24 Items (HAM-D-24) measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 76. The higher the score, the more severe.
Time Frame: Baseline and Week 52
Population: FAS; OC
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Number analyzed (Participants) | 342
units on a scale | -6.86 (8.45)

5. Secondary Outcome: Change From Baseline in HAM-A Total Score After 52 Weeks of Treatment
Description: The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
Time Frame: Baseline and Week 52
Population: FAS; OC
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Number analyzed (Participants) | 342
units on a scale | -5.44 (7.08)

6. Secondary Outcome: Change From Baseline in CGI-S Score After 52 Weeks of Treatment
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
Time Frame: Baseline and Week 52
Population: FAS; OC
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Number analyzed (Participants) | 342
units on a scale | -1.00 (1.22)

7. Secondary Outcome: Proportion of Responders at Week 52 (Response Defined as a >=50% Decrease in MADRS Total Score)
Time Frame: Week 52
Population: FAS; OC; Baseline from lead-in study NCT00635219 / 11984A
Measure: Mean (Standard Deviation); unit: percentage of patients
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Number analyzed (Participants) | 329
percentage of patients | 94.2 (23.4)

8. Secondary Outcome: Proportion of Remitters at Week 52 (Remission Defined as a MADRS Total Score <=10)
Time Frame: Week 52
Population: FAS; OC; Baseline from lead-in study NCT00635219 / 11984A
Measure: Mean (Standard Deviation); unit: percentage of patients
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Number analyzed (Participants) | 329
percentage of patients | 83.0 (37.6)

9. Secondary Outcome: Proportion of Patients With a MADRS Total Score >=22 After 52 Weeks of Treatment
Time Frame: Baseline and Week 52
Population: FAS; OC
Measure: Number; unit: percentage of patients
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Number analyzed (Participants) | 329
percentage of patients | 2.74

10. Secondary Outcome: Change From Baseline in SDS Total Score After 52 Weeks of Treatment
Description: The Sheehan Disability Scale (SDS) comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). The higher the score, the more severe.
Time Frame: Baseline and Week 52
Population: FAS; OC
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Number analyzed (Participants) | 285
units on a scale | -5.60 (6.91)

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 52-week open label period and 4-week safety follow-up period Other Adverse Events: 52-week open label period
Arm/Group | Vortioxetine 2.5, 5, or 10 mg/Day
Serious Adverse Events (participants affected / at risk) | 18/535
Other Adverse Events (participants affected / at risk) | 256/535
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Vortioxetine 2.5, 5, or 10 mg/Day (N=535)
Chest pain (General disorders) | 1
Appendicitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Suicidal ideation (Psychiatric disorders) | 3
Suicide attempt (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1/366
Dermatitis herpetiformis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine 2.5, 5, or 10 mg/Day (N=535)
Nausea (Gastrointestinal disorders) | 106
Influenza (Infections and infestations) | 27
Nasopharyngitis (Infections and infestations) | 56
Accidental overdose (Injury, poisoning and procedural complications) | 29
Weight increased (Investigations) | 31
Dizziness (Nervous system disorders) | 34
Headache (Nervous system disorders) | 82
Insomnia (Psychiatric disorders) | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The main publication has to be published before any sub-publications. H. Lundbeck A/S follows the Vancouver declaration with respect to authorship.